CLINICAL TRIAL: NCT04594148
Title: Triggering Motor Memory Consolidation in Healthy Aging: the Effects of Complex Practice on Brain Activity During Learning of Postural Tasks
Brief Title: The Effect of Training on Brain Activity During Postural Tasks in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Alice Nieuwboer, Full professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S62917
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Healthy Aging
Keywords: Ageing; Motor learning; Postural control; fNIRS; Dual-tasking; Weight-shifting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight-shift training (Experimental): The experimental group will receive a single session of 10x 2.5min of weight-shift training with the VR Wasp Game
  Interventions: Behavioral: Weight-shift training
- Passive control (No Intervention): The passive control group will not receive any form of training. Instead, they will relax for 25min (i.e. talking with the researcher and/or reading a magazine)

INTERVENTIONS:
Behavioral: Weight-shift training — Weight-shift training will consist of a single session of 10x 2.5min of mediolateral weight-shifting in the VR Wasp Game. Including breaks, the session will approximately take 45min.
  Arms: Weight-shift training

SUMMARY:
Older people show deficits in dynamic weight-shifting, as the investigators found that more time is needed to perform weight-shifts and the movements became less fluent and accurate in older versus younger adults. Deficits with weight-shifting in the mediolateral (left-right) direction have been linked to balance and falls in ageing. Balance control can be improved with training. Virtual reality (VR) based training programs for improving balance are gaining ground, as it can provide both fun and challenging balance tasks, enhancing motivation. The investigators demonstrated earlier that older adults show an overloaded neural activation pattern compared to young adults when performing the same VR-based mediolateral weight-shifting task (wasp game). What is yet unclear, is whether improved balance capacity can be gained with training and whether such an intervention impacts the underlying neural mechanisms. Using a combination of behavioral assessments and functional Near-Infrared Spectrocopy (fNIRS), the primary aim of this study is to investigate the effects of a VR-based weight-shift training and its underlying neural imprint in older adults. Furthermore, as a previous study done by the investigators also showed that adding an extra cognitive task in a so-called dual-task (DT) negatively affects weight-shifting performance, a secondary aim will be to test whether weight-shift training will enhance performance during such DT conditions. The results of this study may contribute to the future design of technology-based rehabilitation programs.

DETAILED DESCRIPTION:
For this study, 40 healthy older adults will be included. A previous fNIRS study done by the investigators (unpublished) revealed that our primary outcome, weight-shifting speed, improved from 0,0668 ± 0,0255 m/s to 0,0916 ± 0,0350 m/s. Based on Caljouw et al. (2016), the investigators expect a training effect size of 20%, resulting in a weight-shifting speed of 0.1094 ± 0,0418 m/s. Applying a power of 80% and alpha of 0.05 for a repeated measures ANOVA with a within-between interaction design (within: pre vs post; between: training vs control) the investigators calculated a total sample size of 40 participants (20 per group). Considering possible data exclusion due to fNIRS measurements, the collected fNIRS data will be monitored during recruitment, and more participants will be recruited if necessary.

Prior to training on day 1, participants will be screened for inclusion based on the Montreal Cognitive Assessment (MoCA). Other cognitive assessments include the Flanker (inhibition), Set-Shifting (shifting attention), and Benton Judgement of Line Orientation (visuospatial ability) test, which will be administered on day 2. The Falls Efficacy Scale International (FES-I), a sarcopenia questionnaire (SARC-F), and the Pittsburgh Sleep Quality Index (PSQI) will also be administered on day 2 to assess fear of falling, sarcopenia, and the quality of sleep of the night between day 1 and day 2 of the experiment, respectively.

For both weight-shifting assessment and training, the VR-based Wasp Game will be used. Before starting the Wasp Game, functional limits of stability (fLOS) will be assessed by asking the participant to move the Centre of Mass (CoM) as far as possible over its base of support in eight different directions by pushing a virtual bar away from the center position. Mean CoM shifts will be calculated and used for personalized scaling of the Wasp Game. The Wasp Game was developed and piloted to meet the requirements for balance training for older people and can capture weight-shifting speed and accuracy as learning outcomes. In the Wasp Game, the player is in the middle of an area infested by wasps. By moving the CoM towards a pre-defined 80% of the fLOS, a water stream will come on to hit the wasp. The Wasp Game single-task (WASP-ST) involves hitting wasps in the mediolateral (ML) direction only. During the Wasp Game dual-task (WASP-DT), a serial subtraction task is added as the secondary task, whereby the red ball (representing the CoM) will change color from red to white and white to red within a random interval between 2-5 seconds. A starting number will appear on the screen for 1.5 seconds at the beginning of each trial. Every time the ball changes its color, subtractions have to be made in threes. Subjects will indicate the correct number afterward, so as not to disturb the fNIRS recording.

During training on day 1, participants will perform 10 blocks of 2.5 min weight-shifting within the WASP-ST. Before, and 24h after training, balance performance will be assessed with the Mini Balance Evaluation Systems Test (MiniBEST), and weight-shifting ability with the fLOS, the WASP-ST, and WASP-DT. During the WASP-ST and WASP-DT, oxygenated (HbO2) and deoxygenated hemoglobin (HHb) will be assessed simultaneously by means of functional Near-Infrared Spectroscopy (fNIRS). To be able to compare HbO2 and HHb levels relative to a baseline, both the WASP-ST and WASP-DT will be offered in a block design of 20 sec standing still and looking at a screen capture of the Wasp Game and 20 sec of weight-shifting within the Wasp Game, alternating in 7 trials. Cortical regions assessed with fNIRS include the prefrontal cortex (PFC), frontal eye fields (FEF), premotor cortex (PMC), supplementary motor area (SMA), and supplementary sensory cortex (SSC). To ensure similar fNIRS recording on all test moments, the fNIRS cap and optodes will remain in place between pre and post-testing. Between post and retention testing, certain spots on the head (i.e. Cz) will be marked to guide cap placement on day 2. In a recent study, fNIRS was found to have adequate test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Being able to independently stand upright > 5min

Exclusion Criteria:

* Visual impairment precluding following the targets on the screen
* Cognitive impairment (MoCA<24/26?) / (MMSE<24)?
* History of neurological disorders
* Balance impairments (i.e. vestibular disorders)
* Chronic musculoskeletal, cardiovascular and respiratory conditions
* Diabetes related polyneuropathy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Mediolateral weight-shifting speed | 2 days
  Change in weight-shifting speed during the wasp game in the mediolateral direction from directly before to directly after intervention, from directly before to 24h after intervention and from directly after to 24h after intervention. As weight-shifting tends to slow down when reaching the 80% stability limit to aim for the wasp, mediolateral weight-shifting speed will be determined between 90% of the 80% stability limit on the right side to 90% of the 80% stability limit on the left side and vice versa.

SECONDARY OUTCOMES:
#wasps hit | 2 days
  Change in the number of wasps hit during the wasp game from directly before to directly after intervention, from directly before to 24h after intervention and from directly after to 24h after intervention.
AP trajectory error | 2 days
  Change in the weight-shifting error from the ideal trajectory during the wasp game in the anterior-posterior direction from directly before to directly after intervention, from directly before to 24h after intervention and from directly after to 24h after intervention.
functional limits of stability (fLOS) | 2 days
  Change in the functional limits of stability in eight directions (anterior, anterior-right, right, posterior-right, posterior, posterior-left, left, anterior-right) from directly before to directly after intervention, from directly before to 24h after intervention and from directly after to 24h after intervention.
Oxygenated hemoglobin | 2 days
  Change in oxygenated hemoglobin as measured with functional Near-Infrared Spectroscopy (fNIRS) in five brain regions (prefrontal cortex, frontal eye fields, premotor cortex, supplementary motor area, somatosensory cortex) from directly before to directly after intervention, from directly before to 24h after intervention and from directly after to 24h after intervention.

OTHER OUTCOMES:
Mini Balance Evaluation Systems Test | 2 days
  Change in total Mini Balance Evaluation Systems Test (MiniBEST) score from directly before to 24h after intervention. The MiniBEST is scored on a scale from 0 to 28, where higher scores represent a better outcome.
Deoxygenated hemoglobin | 2 days
  Change in oxygenated hemoglobin as measured with functional Near-Infrared Spectroscopy (fNIRS) in five brain regions (prefrontal cortex, frontal eye fields, premotor cortex, supplementary motor area, somatosensory cortex) from directly before to directly after intervention, from directly before to 24h after intervention and from directly after to 24h after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Nieuwboer, PhD, Principal Investigator — KU Leuven
Locations (1):
- Department of Rehabilitation Sciences KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caljouw SR, Veldkamp R, Lamoth CJ. Implicit and Explicit Learning of a Sequential Postural Weight-Shifting Task in Young and Older Adults. Front Psychol. 2016 May 24;7:733. doi: 10.3389/fpsyg.2016.00733. eCollection 2016. PMID 27252670
- [Background] Willaert J, De Vries AW, Tavernier J, Van Dieen JH, Jonkers I, Verschueren S. Does a novel exergame challenge balance and activate muscles more than existing off-the-shelf exergames? J Neuroeng Rehabil. 2020 Jan 15;17(1):6. doi: 10.1186/s12984-019-0628-3. PMID 31941518

DOCUMENTS (2):
  • Study Protocol (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04594148/Prot_002.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04594148/SAP_003.pdf